CLINICAL TRIAL: NCT04283162
Title: Efficacy of Calcium Dobesilate in Treating Chinese Patients With Mild to Moderate Non-proliferative Diabetic Retinopathy (CALM-DR): a Single-blind, Multicenter, Cluster-randomized, Controlled Trial
Brief Title: Using Calcium Dobesilate to Treat Chinese Patients With Mild to Moderate Non-proliferative Diabetic Retinopathy
Acronym: CALM-DR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Zilin Sun, Chief Physician, Professor of Medicine, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZhongdaH-February
Record Dates: First submitted 2020-02-16; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Retinopathy
Keywords: calcium dobesilate; mild to moderate non-proliferative diabetic retinopathy; cluster-randomized controlled trial
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional treatment plus calcium dobesilate (Experimental): maintain lifestyle habits and the usual treatment, plus the use of calcium dobesilate (500 mg, orally, 3 times per day) for 12 months
  Interventions: Drug: Calcium Dobesilate; Other: conventional treatment
- conventional treatment group (Active Comparator): maintain lifestyle habits and the usual treatment for 12 months
  Interventions: Other: conventional treatment

INTERVENTIONS:
Drug: Calcium Dobesilate — use calcium dobesilate at the dosage of 500 mg, orally, 3 times per day, for 12 months
  Other Names: calcium dobesilate use
  Arms: conventional treatment plus calcium dobesilate
Other: conventional treatment — maintain lifestyle habits and the usual treatment
  Other Names: usual care

SUMMARY:
Calcium dobesilate has been recommended to treat diabetic retinopathy due to its potential in protecting against retinal vascular damage. However, there was limited evidence exploring its efficacy in combating diabetic retinopathy progression. This study, a single-blind, multicenter, cluster-randomized, controlled superiority trial, was designed to evaluate whether calcium dobesilate could prevent diabetic retinopathy progression into an advanced stage among Chinese patients with mild to moderate non-proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
A total of 1,200 patients with mild to moderate non-proliferative diabetic retinopathy will be enrolled and randomly assigned at a ratio of 1:1 into the control group (that is, conventional treatment group) and the intervention group (that is, conventional treatment plus calcium dobesilate [500 mg, 3 times per day] for 12 months). The severity of diabetic retinopathy will be assessed by the Early Treatment Diabetic Retinopathy Study scale.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mild to moderate diabetic retinopathy
* Being older than 18 years
* Being willing to attend this trial.

Exclusion Criteria:

* Being allergic hypersensitive to experimental drugs or comparator drugs
* Having alanine aminotransferase or aspartate aminotransferase ≥2 times higher than the upper limit of normal value, or total bilirubin ≥1.5 times higher than the upper limit of normal value upon the exclusion of mild fatty liver disease
* Having severe renal insufficiency (defined as an estimated glomerular filtration rate ≤30 mL/min/1.73 m^2)
* Having malignant tumor and some other life-threatening diseases
* Being in pregnancy, expecting pregnancy, or breast feeding
* Being with unstable conditions, such as: uncontrolled high blood pressure (e.g., blood pressure >180/100 mmHg); hemoglobin A1c >8.0% or uncontrolled high blood glucose or hypoglycemia; acute cardiovascular events like unstable angina, congestive heart failure, stroke, transient ischemic attack, or myocardial infarction within the previous 3 months; uncontrolled infection; and diabetic ketoacidosis or hyperosmolar state in the past 1 month
* Being with glaucoma, cataracts, or other opacities that may interfere with retinal examination and fundus photography
* Receiving laser treatment, cryo-coagulation, or vitrectomy
* Taking drugs such as diabetic retinopathy or traditional Chinese medicine that may help to improve micro-vascular function in the past 2 weeks
* Receiving vascular endothelial growth factor therapy in the past 4 months or will be judged to take vascular endothelial growth factor therapy because of disease progression
* Having attended other clinical trials in the past 1 month, being attending some clinical trials, or some other conditions that were judged unfit for this trial by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
The rate of the progression of diabetic retinopathy | from baseline to the end of treatment (12 months later)
  Diabetic retinopathy progression is defined as an increase of 2 or more steps on the Early Treatment Diabetic Retinopathy Study scale during follow-up.

SECONDARY OUTCOMES:
Changes in eyesight | 3-month, 6-month, and 12-month from baseline
  Changes in eyesight assessed by visual chart at 4 m by optometrists
Changes in the numbers, location, and types of the retinal lesions | 3-month, 6-month, and 12-month from baseline
  Using retinal photography to detect the changes in the numbers, location, and types of the retinal lesions at different time-points
Changes in the retinal blood vessel diameter and arteriovenous ratio | 3-month, 6-month, and 12-month from baseline
  Using photography (optic disc-centered photograph) to detect the retinal blood vessel diameter and arteriovenous ratio at different time-points
Changes in metabolic biomarkers such as HbA1c | 3-month, 6-month, and 12-month from baseline
  The metabolic biomarkers were assessed by laboratory measurement at different time-points

CONTACTS AND LOCATIONS:
Overall Officials: Zilin Sun, Ph.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Department of Endocrinology, Zhongda Hospital, Institute of Diabetes, Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Hu H, Liu J, Wang D, Qiu S, Yuan Y, Wang F, Wen L, Song Q, Sun ZL. Efficacy of calcium dobesilate in treating Chinese patients with mild-to-moderate non-proliferative diabetic retinopathy (CALM-DR): protocol for a single-blind, multicentre, 24-armed cluster-randomised, controlled trial. BMJ Open. 2021 May 28;11(5):e045256. doi: 10.1136/bmjopen-2020-045256. PMID 34049911